CLINICAL TRIAL: NCT05429827
Title: The Therapeutic Effects of Dextrose Injection for Myofascial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ta-Shen Kuan, MD, associate professor, M.D., National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-BR-110-078
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Myofascial Trigger Point Pain
Keywords: myofascial trigger point; endplate noise; dextrose.
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Saline Solution; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal saline (Placebo Comparator): Injection of 2 ml normal saline into a myofascial trigger point.
  Interventions: Other: normal saline
- hypo-osmolar dextrose solution (Experimental): Injection of 2 ml 5% dextrose into a myofascial trigger point.
  Interventions: Drug: Dextrose 5% in water
- hyper-osmolar dextrose solution (Experimental): Injection of 2 ml 15% dextrose into a myofascial trigger point.
  Interventions: Drug: Dextrose 15% in water

INTERVENTIONS:
Other: normal saline — Inject 2 ml normal saline into a myofascial trigger point and evaluate the clinical effects before and after the injection.
  Arms: Normal saline
Drug: Dextrose 5% in water — Inject 2 ml 5% dextrose into a myofascial trigger point and evaluate the clinical effects before and after the injection.
  Arms: hypo-osmolar dextrose solution
Drug: Dextrose 15% in water — Inject 2 ml 15% dextrose into a myofascial trigger point and evaluate the clinical effects before and after the injection.
  Arms: hyper-osmolar dextrose solution

SUMMARY:
Patients with an myofascial trigger point (MTrP) in their upper trapezius will be divided into three groups: Group A receiving MTrP injection with normal saline (control group), Group B with hypo-osmolar dextrose (5% dextrose), and Group C with hyper-osmolar dextrose (15% dextrose). Clinical outcomes and morphological changes will be measured before the injection, one hour after, one week after, two weeks after, and one month after the injection to delineate the therapeutic effects of dextrose injection for an MTrP.

DETAILED DESCRIPTION:
This experiment is designed to evaluate the therapeutic effects of dextrose injection on an myofascial trigger point (MTrP). Patients with an MTrP in their upper trapezius will be recruited and be divided into three groups: Group A receiving MTrP injection with normal saline (control group), Group B with hypo-osmolar dextrose (5% dextrose), and Group C with hyper-osmolar dextrose (15% dextrose). Clinical outcomes (visual analog scale, pressure pain threshold, range of motion, neck disability index) will be measured before the injection, one hour after, one week after, two weeks after, and one month after the injection. Morphological changes of an MTrP before, and after the injection will also be evaluated by sonography. Through this study, the definite therapeutic effects, and the better osmolality of dextrose injection for the treatment of an MTrP will be delineated.

ELIGIBILITY:
Inclusion Criteria:

* 1). Patients should be 20 years of age or older;
* 2). They are able to communicate freely;
* 3). Patients have the diagnosis of myofascial pain syndrome (MPS) with a definite myofascial trigger point (MTrP) in the neck base and upper back regions (the upper trapezius muscle). The MTrP is identiﬁed based on the following criteria, as recommended by Simons [Simons et al., 1999]:

  * (a). a localized tender spot in a palpable taut band of muscle ﬁbers,
  * (b). recognized pain (as the usual clinical complaint) when the tender spot is compressed,
  * (c). characteristic and consistent referred pain.
* 4). Symptoms of MPS should be more than 3 weeks.

Exclusion Criteria:

* (1). acute or serious medical problems;
* (2). cognitive impairment or psychiatric disorder;
* (3). coagulopathy or any other bleeding disorder;
* (4). taking medication of anticoagulation or antithrombolytics;
* (5). sensory deficiency over the body part where MTrPs located;
* (6). serum hepatitis B or acquired immunodeﬁciency syndrome;
* (7). malignancy;
* (8). pregnant or likely to be pregnant.
* (9). diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) | Change from Baseline visual analog scale at one hour after intervention.
  To measure the pain intensity of a myofascial trigger point. The minimum value is 0, and the maximum value is 10, and higher scores mean worse outcome (more painful).
visual analog scale (VAS) | Change from Baseline visual analog scale at one week after intervention.
  To measure the pain intensity of a myofascial trigger point. The minimum value is 0, and the maximum value is 10, and higher scores mean worse outcome (more painful).
visual analog scale (VAS) | Change from Baseline visual analog scale at two weeks after intervention.
  To measure the pain intensity of a myofascial trigger point. The minimum value is 0, and the maximum value is 10, and higher scores mean worse outcome (more painful).
visual analog scale (VAS) | Change from Baseline visual analog scale at one month after intervention.
  To measure the pain intensity of a myofascial trigger point. The minimum value is 0, and the maximum value is 10, and higher scores mean worse outcome (more painful).

SECONDARY OUTCOMES:
pressure pain threshold (PPT) | Change from Baseline pressure pain threshold at one hour after intervention.
  To measure the change of pressure pain threshold of a myofascial trigger point. The minimum value is 0 Kg/cm2, the maximum value is 5 Kg/cm2, and higher scores mean better outcome (less painful).
pressure pain threshold (PPT) | Change from Baseline pressure pain threshold at one week after intervention.
  To measure the change of pressure pain threshold of a myofascial trigger point. The minimum value is 0 Kg/cm2, the maximum value is 5 Kg/cm2, and higher scores mean better outcome (less painful).
pressure pain threshold (PPT) | Change from Baseline pressure pain threshold at two weeks after intervention.
  To measure the change of pressure pain threshold of a myofascial trigger point. The minimum value is 0 Kg/cm2, the maximum value is 5 Kg/cm2, and higher scores mean better outcome (less painful).
pressure pain threshold (PPT) | Change from Baseline pressure pain threshold at one month after intervention.
  To measure the change of pressure pain threshold of a myofascial trigger point. The minimum value is 0 Kg/cm2, the maximum value is 5 Kg/cm2, and higher scores mean better outcome (less painful).
Range of motion (ROM) of the neck | Change from Baseline range of motion (ROM) of the neck at one hour after intervention.
  To measure the change of the range of motion of cervical spine. The minimum value is 0 degree, the maximum value is 90 degree, and higher scores mean better outcome.
Range of motion (ROM) of the neck | Change from Baseline range of motion (ROM) of the neck at one week after intervention.
  To measure the change of the range of motion of cervical spine. The minimum value is 0 degree, the maximum value is 90 degree, and higher scores mean better outcome.
Range of motion (ROM) of the neck | Change from Baseline range of motion (ROM) of the neck at two weeks after intervention.
  To measure the change of the range of motion of cervical spine. The minimum value is 0 degree, the maximum value is 90 degree, and higher scores mean better outcome.
Range of motion (ROM) of the neck | Change from Baseline range of motion (ROM) of the neck at one month after intervention.
  To measure the change of the range of motion of cervical spine. The minimum value is 0 degree, the maximum value is 90 degree, and higher scores mean better outcome.
neck disability index (NDI) | Change from Baseline neck disability index (NDI) at one hour after intervention.
  To measure the change of neck disability index (NDI) related to the myofascial trigger point. The minimum value is 0, the maximum value is 50, and higher scores mean worse outcome (increased functional disability).
neck disability index (NDI) | Change from Baseline neck disability index (NDI) at one week after intervention.
  To measure the change of neck disability index (NDI) related to the myofascial trigger point. The minimum value is 0, the maximum value is 50, and higher scores mean worse outcome (increased functional disability).
neck disability index (NDI) | Change from Baseline neck disability index (NDI) at two weeks after intervention.
  To measure the change of neck disability index (NDI) related to the myofascial trigger point. The minimum value is 0, the maximum value is 50, and higher scores mean worse outcome (increased functional disability).
neck disability index (NDI) | Change from Baseline neck disability index (NDI) at one month after intervention.
  To measure the change of neck disability index (NDI) related to the myofascial trigger point. The minimum value is 0, the maximum value is 50, and higher scores mean worse outcome (increased functional disability).

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Shen Kuan, M.D., M.S., Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Department of physical Medicine and Rehabilitation, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou Y, Chiou HJ, Wang HK, Lai YC. Ultrasound-guided dextrose injection treatment for chronic myofascial pain syndrome: A retrospective case series. J Chin Med Assoc. 2020 Sep;83(9):876-879. doi: 10.1097/JCMA.0000000000000339. PMID 32349034
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Hong CZ. Treatment of myofascial pain syndrome. Curr Pain Headache Rep. 2006 Oct;10(5):345-9. doi: 10.1007/s11916-006-0058-3. PMID 16945250
- [Background] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Background] Kuan TS, Chen JT, Chen SM, Chien CH, Hong CZ. Effect of botulinum toxin on endplate noise in myofascial trigger spots of rabbit skeletal muscle. Am J Phys Med Rehabil. 2002 Jul;81(7):512-20; quiz 521-3. doi: 10.1097/00002060-200207000-00008. PMID 12131178